CLINICAL TRIAL: NCT03640832
Title: A Clinical Study to Assess the Local Cutaneous and Ocular Tolerance of a Developmental Cosmetic Facial Serum Formulation in Healthy Females With Sensitive Skin
Brief Title: A Clinical Study to Investigate the Dermal and Ocular Tolerance of a Developmental Cosmetic Facial Serum Formulation in Healthy Females With Sensitive Skin
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 209442
Record Dates: First submitted 2018-08-17; First posted 2018-08-21 (Actual); Results first posted 2019-10-01 (Actual); Last update posted 2020-11-27 (Actual); Status verified 2020-11

CONDITIONS: Skin Care

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Evaluator blinded (dermatologist and ophthalmologist).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Test product (Experimental): All the participant in this arm will receive the test product (development serum). Test product will be applied twice daily to the freshly cleansed skin in place of the participant's current serum and before applying moisturizer.
  Interventions: Other: Developmental Serum
- Reference product (Active Comparator): All the participant in this arm will receive the reference product (Physiogel Calming Relief Anti-Redness Serum). Reference product will be applied twice daily to the freshly cleansed skin in place of the participant's current serum and before applying moisturizer.
  Interventions: Other: Physiogel Calming Relief Anti-Redness Serum

INTERVENTIONS:
Other: Developmental Serum — A 30millilitre (mL) bottle with a piston pump will be dispensed to the participants, to be used as a topical dermal (facial) application, twice daily as per normal home use.
  Arms: Test product
Other: Physiogel Calming Relief Anti-Redness Serum — A 30mL bottle with a piston pump will be dispensed to the participants, to be used as a topical dermal (facial) application, twice daily as per normal home use.
  Arms: Reference product

SUMMARY:
To determine the local cutaneous and ocular tolerance of a developmental cosmetic facial serum in healthy females with sensitive facial skin under normal conditions of use.

DETAILED DESCRIPTION:
This is a single-center, non-comparative clinical 'in-use' study to determine the local cutaneous and ocular tolerance of a developmental cosmetic facial serum formulation in healthy female subjects aged 18 to 65 years (inclusive) with clinically evaluated sensitive skin, as determined by a positive response to a Lactic Acid Sting Test (LAST), with minimal signs or symptoms of cutaneous irritation and no signs or symptoms of ocular irritation. A reference product, proven to be suitable for use in a sensitive skin population will also be used.

ELIGIBILITY:
Inclusion Criteria:

* Subject provision of a signed and dated informed consent document indicating that the subject has been informed of all pertinent aspects of the study before any assessment is performed.
* A subject who is willing and able to comply with scheduled visits, the application schedule, the lifestyle guidelines, and other study procedures.
* A subject in good general and mental health with, in the opinion of the investigator or medically qualified designee (if the investigator is not suitably qualified), no clinically significant/relevant abnormalities in medical history or upon dermatologist and ophthalmologist examination, or condition, that would impact the subject's safety, wellbeing or the outcome of the study, if they were to participate in the study, or affect the individual's ability to understand and follow study procedures and requirements.
* A subject with sensitive facial skin, defined as a positive response to a lactic acid sting test in the nasolabial area.
* A subject with a dermatologist signs and symptoms of cutaneous irritation score of greater than or equal to 0.5 (very slight) for erythema.
* A subject with a dermatologist signs and symptoms of cutaneous irritation score of greater than or equal to 0.5 (very slight) for dryness.
* A subject with a dermatologist signs and symptoms of cutaneous irritation score of 0 (none) or 0.5 (very sight) for scaling.
* A subject with a dermatologist signs and symptoms of cutaneous irritation score of 0 (none) or 0.5 (very sight) for edema.
* A subject with an ophthalmologist total signs and symptoms of ocular irritation score of 0 (none).

Exclusion Criteria:

* A subject who is an employee of the investigational site, either directly involved in the conduct of the study or a member of their immediate family; or an employee of the investigational site otherwise supervised by the investigator; or, a GSK CH employee directly involved in the conduct of the study or a member of their immediate family.
* A subject who has participated in other studies (including non-medicinal studies) involving investigational product(s) within 30 days prior to study entry and/or during study participation.
* A subject with, in the opinion of the investigator or medically qualified designee, an acute or chronic medical or psychiatric condition that may increase the risk associated with study participation or investigational product administration or may interfere with the interpretation of study results and, in the judgment of the investigator or medically qualified designee, would make the subject inappropriate for entry into this study.
* A subject who is pregnant (self-reported).
* A subject who is breastfeeding.
* A subject with known or suspected intolerance or hypersensitivity to the study materials (or closely related compounds) or any of their stated ingredients.
* A subject who, in the opinion of the investigator or medically qualified designee, should not participate in the study.
* A subject unwilling or unable to comply with the Lifestyle Considerations required by this study, as described in this protocol.
* A subject with current or recent (within last 6 months before the start of the study) history of atopic lesions and/or eczema.
* A subject with a history of allergic reactions to topical-use products, cosmetics or medications or their ingredients.
* A subject with any history of significant diseases or medical conditions known to alter skin or eye appearance or physiologic response (e.g. diabetes) which could, in the opinion of the Investigator, preclude topical application of the investigational products and/or interfere with the evaluation of the test site reaction.
* A subject presenting open sores, pimples, or cysts at the application site (face).
* A subject with an active dermatosis (local or disseminated) that might interfere with the results of the study.
* A subject with a dermatologist signs and symptoms of cutaneous irritation score of 3 (severe) for erythema, edema, scaling or dryness.
* A subject considered immune-compromised.
* A subject currently using any medication which in the opinion of the investigator, may affect the evaluation of the investigational product, or place the subject at undue risk.
* A subject who has used any of the following topical or systemic medications up to two weeks before the screening visit: immuno-suppressants, antihistamines, non-steroidal anti-inflammatory drugs (NSAIDS), and/or corticosteroids.
* A subject who has used oral or topical treatment with vitamin A acid and/or its derivatives up to 1 month before the screening visit.
* A subject who has been vaccinated up to 1 month before the screening visit or who are intending to receive a vaccination during their participation in the study.
* A subject with a recent history (within the last 5 years) of alcohol or other substance abuse.
* A subject with any skin marks on the face that might interfere with the evaluation of possible skin reactions (e.g. pigmentation disorders, vascular malformations, scars, tattoos, excessive hair, numerous freckles).
* Subjects with corneal ulcers, keratoconus, blepharitis, meibomitis, pterygium, chemosis,moderately or severe hyperemia or other active ocular diseases.
* A subject who has previously been enrolled in this study.

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Female who, at the time of screening, is between the ages of 18 and 65 years, inclusive.
Enrollment: 90 (Actual)
Dates: Start 2018-10-15 (Actual); Primary Completion 2018-11-13 (Actual); Study Completion 2018-11-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Schenefeld, Schleswig-Holstein, Germany

IPD SHARING:
Plan to Share IPD: Yes
IPD for this study is available via the Clinical Study Data Request site.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD is available via the Clinical Study Data Request site (copy the URL below to your browser)
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months.
URL: https://www.clinicalstudydatarequest.com/Posting.aspx?ID=20740

RESULTS

PARTICIPANT FLOW:
Recruitment Details: All the participants were enrolled from one center in Germany.
Pre-assignment Details: A total of 141 participants were screened for the study out of which 90 participants were enrolled and randomized to any of the 2 treatment arms. A total of 51 participants did not meet the study criteria and were not randomized. All 90 randomized participants completed the study.
Groups:
- Developmental Facial Serum (Test Product): Participants were randomized to topically (facial) apply Physiogel Developmental Facial Serum, twice daily (morning and evening) to the freshly cleansed skin before applying moisturizer up to 21 (+2) days
- Physiogel Calming Relief Anti-redness Serum(Reference Product): Participants were randomized to topically (facial) apply Physiogel Calming Relief Anti-Redness Serum, twice daily (morning and evening) to the freshly cleansed skin before applying moisturizer up to 21 (+2) days
Period: Overall Study
Arm/Group | Developmental Facial Serum (Test Product) | Physiogel Calming Relief Anti-redness Serum(Reference Product)
Started | 44 | 46
Completed | 44 | 46
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: The Safety Population included all participants who received at least 1 dose of the study product (test or reference product).
Groups:
- Total: Total of all reporting groups
Arm/Group | Developmental Facial Serum (Test Product) | Physiogel Calming Relief Anti-redness Serum(Reference Product) | Total
Number analyzed (Participants) | 44 | 46 | 90
Age, Continuous [Mean (Standard Deviation); unit: Years] | 49.5 (10.05) | 48.8 (11.84) | 49.2 (10.95)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 44 | 46 | 90
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian - South East Asian heritage | 0 | 1 | 1
  White - White/Caucasian/European heritage | 43 | 44 | 87
  Unknown or not reported | 1 | 1 | 2
Fitzpatrick Skin Type [Count of Participants; unit: Participants]
  I - pale white skin | 6 | 4 | 10
  II - white skin | 13 | 23 | 36
  III - light brown skin | 22 | 17 | 39
  IV - moderate brown skin | 3 | 2 | 5
Dermatologist Assessment of Signs and Symptoms of Cutaneous Irritation Total Score at Baseline [Count of Participants; unit: Participants] — A qualified dermatologist visually assessed the signs and symptoms of cutaneous irritation for dermal erythema, dryness, scaling, and edema on a scale with a score range of 0 to 3, where 0=none, 0.5=very slight, 1=slight, 2=moderate, 3=severe. Cutaneous irritation total score = dermal score of erythema + dermal score of dryness + dermal score of scaling + dermal score of edema. Total possible score range is 0 to 12 (higher value indicated more cutaneous irritation).
  Participants
    Baseline, total score(TS)= 1 | 11 | 14 | 25
    Baseline, TS= 1.5 | 16 | 12 | 28
    Baseline, TS= 2 | 7 | 3 | 10
    Baseline, TS= 2.5 | 1 | 6 | 7
    Baseline, TS= 3 | 5 | 6 | 11
    Baseline, TS= 3.5 | 1 | 1 | 2
    Baseline, TS= 4 | 2 | 4 | 6
    Baseline, TS= 4.5 | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With a Unit Change of Greater Than (>) 1 in Signs and Symptoms of Cutaneous Irritation Total Scores From Baseline to 21 Days of Product Use
Description: A qualified dermatologist visually assessed the signs and symptoms of cutaneous irritation for dermal erythema, dryness, scaling, and edema on a scale with a score range of 0 to 3, where 0=none, 0.5=very slight, 1=slight, 2=moderate, 3=severe. Cutaneous irritation total score = dermal score of erythema + dermal score of dryness + dermal score of scaling + dermal score of edema. Total possible score range is 0 to 12 (higher value indicated more cutaneous irritation). Change from baseline for 21 days of product use = total score at Day 21 minus total score at baseline. Participants with a unit change of greater than (>) 1 in total score (TS) of cutaneous irritation from baseline to 21 days of product use, are reported in this outcome measure.
Time Frame: Baseline and Day 21
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Developmental Facial Serum (Test Product) | Physiogel Calming Relief Anti-redness Serum(Reference Product)
Number analyzed (Participants) | 44 | 46
Participants | 3 | 0

2. Secondary Outcome: Number of Participants With a Unit Change of >1 in Signs and Symptoms of Ocular Irritation Total Scores From Baseline to 21 Days of Product Use
Description: A qualified ophthalmologist visually assessed the signs and symptoms of ocular irritation for ocular eczema of the eyelid, conjunctivitis, follicles and chemosis conjunctivae on a scale with a score range of 0 to 3, where 0=none, 0.5=very slight, 1=slight, 2=moderate, 3=severe. Ocular irritation total score = ocular score of eczema of the eyelid + ocular score of conjunctivitis + ocular score of follicles + ocular score of chemosis conjunctivae. Total possible score range is 0 to 12 (higher value indicated more ocular irritation). Change from baseline for 21 days of product use = total score at Day 21 minus total score at baseline. Participants with a unit change of > 1 in total score of ocular irritation from baseline to 21 days of product use, are reported in this outcome measure.
Time Frame: Baseline and Day 21
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Developmental Facial Serum (Test Product) | Physiogel Calming Relief Anti-redness Serum(Reference Product)
Number analyzed (Participants) | 44 | 46
Participants
  Baseline, TS= 0 | 44 | 46
  Change at Day 21, TS >1 | 1 | 0

3. Secondary Outcome: Number of Participants With a Unit Change of >1 in Signs and Symptoms of Cutaneous Irritation (Self-assessment) From Baseline to 1 to 2 Hours Post First Product Use and 21 Days of Product Use
Description: Participants were instructed to self-assess any sensations of cutaneous discomfort for redness, dryness, stinging/burning, itching and tightness on a scale with a score range of 0 to 3, where 0=none, 0.5=very slight, 1=slight, 2=moderate, 3=severe. Participant self-assessment of cutaneous irritation total score = redness + dryness + itching + stinging/burning + tightness. Total possible score range is 0 to 15 (higher value indicated more cutaneous irritation). Change from baseline at 1-2 hours post first use = total score at 1 to 2 hours minus total score at baseline. Similarly, change from baseline for 21 days of product use = total score at Day 21 minus total score at baseline. Participants with a unit change of >1 in total score of cutaneous irritation from baseline to 1-2 hours post first product use and 21 days of product use, are reported in this outcome measure.
Time Frame: Baseline, 1-2 hours post first use, Day 21
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Developmental Facial Serum (Test Product) | Physiogel Calming Relief Anti-redness Serum(Reference Product)
Number analyzed (Participants) | 44 | 46
Participants
  Baseline, TS= 1 | 3 | 1
  Baseline, TS= 1.5 | 1 | 4
  Baseline, TS= 2 | 3 | 4
  Baseline, TS= 2.5 | 2 | 6
  Baseline, TS= 3 | 8 | 2
  Baseline, TS= 3.5 | 1 | 3
  Baseline, TS= 4 | 6 | 9
  Baseline, TS= 4.5 | 4 | 3
  Baseline, TS= 5 | 5 | 4
  Baseline, TS= 5.5 | 1 | 0
  Baseline, TS= 6 | 3 | 2
  Baseline, TS= 6.5 | 0 | 2
  Baseline, TS= 7 | 0 | 2
  Baseline, TS= 7.5 | 1 | 0
  Baseline, TS= 8 | 1 | 3
  Baseline, TS= 9 | 2 | 1
  Baseline, TS= 10 | 2 | 0
  Baseline, TS= 12 | 1 | 0
  Change at 1-2 hours, TS >1 | 3 | 4
  Change at Day 21, TS >1 | 3 | 1

4. Secondary Outcome: Number of Participants With a Unit Change of >1 in Signs and Symptoms of Ocular Irritation (Self-assessment) From Baseline to 1 to 2 Hours Post First Product Use and 21 Days of Product Use
Description: Participants were instructed to self-assess any sensations of ocular discomfort for redness, dryness, stinging/burning and itching on a scale with a score range of 0 to 3, where 0=none, 0.5=very slight, 1=slight, 2=moderate, 3=severe. Participant self-assessment of ocular irritation total score = redness + dryness + itching + stinging/burning. Total possible score range is 0 to 12 (higher value indicated more ocular irritation). Change from baseline at 1-2 hours post first use = total score at 1 to 2 hours minus total score at baseline. Similarly, change from baseline for 21 days of product use = total score at Day 21 minus total score at baseline. Participants with a change of > 1 in total score of ocular irritation from baseline to 1-2 hours post first product use and Day 21 days of product use, are reported in this outcome measure.
Time Frame: Baseline, 1-2 hours post first use, Day 21
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Developmental Facial Serum (Test Product) | Physiogel Calming Relief Anti-redness Serum(Reference Product)
Number analyzed (Participants) | 44 | 46
Participants
  Baseline, TS= 0 | 23 | 22
  Baseline, TS= 0.5 | 10 | 6
  Baseline, TS= 1 | 3 | 8
  Baseline, TS= 1.5 | 4 | 5
  Baseline, TS= 2 | 1 | 3
  Baseline, TS= 2.5 | 1 | 1
  Baseline, TS= 4 | 1 | 0
  Baseline, TS= 6 | 1 | 0
  Baseline, TS= 6.5 | 0 | 1
  Change at 1-2 hours, TS >1 | 0 | 0
  Change at Day 21, TS >1 | 1 | 1

ADVERSE EVENTS:
Time Frame: up to 21 (+2) days
Description: The Safety Population included all participants who received at least 1 dose of the study product (test or reference product). Treatment-emergent adverse events (TEAEs) were defined as new adverse events (AEs) that occurred on or after the first product application. One participant might have experienced more than one AE during the study. All treatment emergent AEs and serious adverse events (SAEs) were collected and reported.
Arm/Group | Developmental Facial Serum (Test Product) | Physiogel Calming Relief Anti-redness Serum(Reference Product)
All-Cause Mortality (participants affected / at risk) | 0/44 | 0/46
Serious Adverse Events (participants affected / at risk) | 0/44 | 0/46
Other Adverse Events (participants affected / at risk) | 10/44 | 7/46
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Developmental Facial Serum (Test Product) (N=44) | Physiogel Calming Relief Anti-redness Serum(Reference Product) (N=46)
Chalazion (Eye disorders) | 0 | 1
Eye paraesthesia (Eye disorders) | 0 | 1
Eye pruritus (Eye disorders) | 1 | 0
Nasopharyngitis (Infections and infestations) | 3 | 0
Arthropod bite (Injury, poisoning and procedural complications) | 1 | 0
Jaw cyst (Musculoskeletal and connective tissue disorders) | 0 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Headache (Nervous system disorders) | 0 | 3
Dysmenorrhoea (Reproductive system and breast disorders) | 1 | 0
Nasal discomfort (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Acne (Skin and subcutaneous tissue disorders) | 3 | 1
Rash macular (Skin and subcutaneous tissue disorders) | 0 | 1
Skin burning sensation (Skin and subcutaneous tissue disorders) | 0 | 1
Skin irritation (Skin and subcutaneous tissue disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Study Protocol (2018-06-13): https://cdn.clinicaltrials.gov/large-docs/32/NCT03640832/Prot_000.pdf
  • Statistical Analysis Plan (2018-09-21): https://cdn.clinicaltrials.gov/large-docs/32/NCT03640832/SAP_001.pdf